CLINICAL TRIAL: NCT07366762
Title: Comparison Between the Effect of Periurethral Injection of Platelet-rich Plasma VS Platelet Rich Fibrin in Treatment of Female Stress Urinary Incontinence
Brief Title: Comparison Between Two Techniques in Treatment of Female Stress Urinary Incontinence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Marwa Reda Mohamed Gebril, obstetrics and gynecology resident, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KFSIRB200-320
Record Dates: First submitted 2026-01-08; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Female Stress Urinary Incontinence
Keywords: PRP- i-PRF- SUI

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group one who had received PRP injections (Active Comparator)
  Interventions: Biological: Platelet Rich Plasma
- group two who had received i-PRF injections (Active Comparator)
  Interventions: Biological: Platelet rich fibrin

INTERVENTIONS:
Biological: Platelet Rich Plasma — Approximately 5 mL of PRP will be injected at three points (on both sides of the urethra and urethrovaginal space) under local anesthesia. Injections will be performed by gynecologist in the outpatient clinic.
  Arms: group one who had received PRP injections
Biological: Platelet rich fibrin — Approximately 5 mL of i-PRF will be injected at three points (on both sides of the urethra and urethrovaginal space) under local anesthesia. Injections will be performed by gynecologist in the outpatient clinic
  Arms: group two who had received i-PRF injections

SUMMARY:
compare the therapeutic effect of periurethral injection of autologous platelet-rich plasma (PRP) and injectable platelet rich fibrin (i-PRF) in treatment of female stress urinary incontinence and comparing the need for re-injection in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with primary symptoms of SUI confirmed by patient's medical history and clinical examination, including a focused incontinence evaluation

  * Age range of 30-75 years
  * Females unfit for surgery
  * Females with SUI recurrence after previous surgical procedure by suburethal sling
  * Females refusing surgical interventions

Exclusion Criteria:

* Residual urine volume exceeding 100 cc after excretion
* Evidence of detrusor over-activity on the urodynamic test
* Active urinary tract or vaginal infection
* Malignancies of the genitourinary system
* Patients with genitourinary fistula or urethral diverticulum

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — stress urinary incontinence in females
Enrollment: 40 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2026-01-02 (Actual)

PRIMARY OUTCOMES:
changes in the severity of SUI measured by Incontinence Impact Questionnaire (IIQ7) | baseline and three and six months follow up

SECONDARY OUTCOMES:
changes in the severity of SUI using 10 point visual analogue scale | baseline and three and six months follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Kafr Elsheikh University Hospital, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: Undecided